CLINICAL TRIAL: NCT00204490
Title: Mammographic Density and Soy Isoflavones
Brief Title: Soy Isoflavones and Breast Cancer Risk Reduction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 03-260; UTMB GCRC #635 (Other: UTMB ITSCRC); R01CA095545 (NIH); M01RR000073 (NIH); 1UL1RR029876-01 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Results first posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer
Keywords: soy; isoflavones; phytoestrogens; prevention; mammographic density; bone density
MeSH Terms: conditions — Breast Neoplasms | interventions — Isoflavones; Carbohydrates; Sugars

STUDY DESIGN:
Intervention Model Description: One group received soy isoflavones (60 mg daidzein, 60 mg gensitein and 16.6 mg glycitein, all as aglycone equivalent) Another group, carbohydrate filler
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Research pharmacist dispensed study pills according to a pre-generated randomization list and were blinded to all other aspects of the study protocol.
  Subjects, research staff, investigators, and statistician all were blinded to treatment assignment.
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): soy isoflavones
  Interventions: Dietary Supplement: isoflavones
- 2 (Placebo Comparator): carbohydrates (maltodextrin)
  Interventions: Dietary Supplement: carbohydrate

INTERVENTIONS:
Dietary Supplement: isoflavones — soy isoflavones: Each tablet contains 246 mg Novasoy, 676 mg calcium, 15 mg riboflavin, and other innert materials to a total weight of 1000 mg. Subject takes two isoflavone tablets plus 1 multi-vitamin per day for five days per week for upto 2 years.
  Other Names: Isoflavone pill
  Arms: 1
Dietary Supplement: carbohydrate — carbohydrate: 246 mg maltodextrin, 676 mg calcium, 15 mg riboflavin and other innert ingredients to a total weight of 1000 mg per tablet. subject takes two tablets plus one multivitamin per day for five days per week for upto 2 years.
  Other Names: Sugar pill
  Arms: 2

SUMMARY:
Soy consumption has been associated with reduced risk for developing breast cancer. Soy contains isoflavones which are weak estrogens. The roles of soy isoflavones in reducing breast cancer risk are currently unclear. Breast density has been considered as a breast cancer risk marker. We hypothesize that because isoflavones have estrogen-like activities, breast density and possibly bone density will be lower in women on soy-isoflavones.

DETAILED DESCRIPTION:
This is a randomized, double-blind study, with two arms and 100 women in each arm. Premenopausal women will be recruited and randomly allocated to take one of the two different dietary supplements in pills daily for 2 years. The two supplements are soy isoflavones (treatment) and placebo (carbohydrates). Both treatment and placebo pills will contain multi-vitamins and minerals. Multiple blood, urine, and breast fluid samples will be obtained before and during the dietary supplement periods and analyzed for biomarkers of breast cancer risk. At baseline and after the intervention period, breast density and bone density will be assessed by radiologic techniques. The efficacy of the dietary intervention will be determined by comparing mean changes of serum markers for breast cancer risk,dense breast tissue, and bone mineral density over the two year dietary intervention period in the two supplement groups with adjustment for baseline values and individual patient characteristics of interest. We predict that 2 years of soy isoflavone supplement will reduce breast density, which may be explained by individual changes in serum markers of breast cancer risk.

ELIGIBILITY:
Inclusion Criteria:

* healthy premenopausal women
* 30 to 42 years old
* normal mammograms
* regular menstrual cycles

Exclusion Criteria:

* abnormal mammograms
* first degree relatives with breast cancer
* pregnant or lactating
* peri- or post-menopause
* breast augmentation, reduction or lifting
* on oral contraceptive medications or exogenous hormones
* medically prescribed diets
* allergic reaction to soy products

Ages: 30 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 197 (Actual)
Dates: Start 2004-04 (Actual); Primary Completion 2012-12-10 (Actual); Study Completion 2023-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee-Jane W Lu, Ph.D., Principal Investigator — The University of Teas Medical Branch
Locations (1):
- General Clinical Reserach Center, The University of Texas Medical Branch, Galveston, Texas, United States

REFERENCES:
- [Derived] Lu LW, Chen NW, Brunder DG, Nayeem F, Nagamani M, Nishino TK, Anderson KE, Khamapirad T. Soy isoflavones decrease fibroglandular breast tissue measured by magnetic resonance imaging in premenopausal women: A 2-year randomized double-blind placebo controlled clinical trial. Clin Nutr ESPEN. 2022 Dec;52:158-168. doi: 10.1016/j.clnesp.2022.10.007. Epub 2022 Oct 26. PMID 36513449
- [Derived] Lu LW, Chen NW, Nayeem F, Nagamani M, Anderson KE. Soy isoflavones interact with calcium and contribute to blood pressure homeostasis in women: a randomized, double-blind, placebo controlled trial. Eur J Nutr. 2020 Sep;59(6):2369-2381. doi: 10.1007/s00394-019-02085-3. Epub 2019 Sep 18. PMID 31535213
- [Derived] Lu LW, Chen NW, Nayeem F, Ramanujam VS, Kuo YF, Brunder DG, Nagamani M, Anderson KE. Novel effects of phytoestrogenic soy isoflavones on serum calcium and chloride in premenopausal women: A 2-year double-blind, randomized, placebo-controlled study. Clin Nutr. 2018 Dec;37(6 Pt A):1862-1870. doi: 10.1016/j.clnu.2017.11.002. Epub 2017 Nov 11. PMID 29183775
- [Derived] Lu LJ, Nishino TK, Johnson RF, Nayeem F, Brunder DG, Ju H, Leonard MH, Grady JJ, Khamapirad T. Comparison of breast tissue measurements using magnetic resonance imaging, digital mammography and a mathematical algorithm. Phys Med Biol. 2012 Nov 7;57(21):6903-27. doi: 10.1088/0031-9155/57/21/6903. Epub 2012 Oct 9. PMID 23044556

RESULTS

PARTICIPANT FLOW:
Groups:
- Soy Isoflavones: Each tablet contains 246 mg Novasoy, 676 mg calcium, 15 mg riboflavin, and other inert materials to a total weight of 1000 mg. Subject takes two isoflavone tablets plus 1 multi-vitamin per day for five days per week for up to 2 years.
- Placebo: Carbohydrate: 246 mg maltodextrin, 676 mg calcium, 15 mg riboflavin and other inert ingredients to a total weight of 1000 mg per tablet. subject takes two tablets plus one multivitamin per day for five days per week for up to 2 years.
Period: Enrollment/Allocation of Qualified Women
Arm/Group | Soy Isoflavones | Placebo
Started | 99 | 98
Completed | 99 | 98
Not Completed | 0 | 0
Period: Follow-up <1 Year
Arm/Group | Soy Isoflavones | Placebo
Started | 99 | 98
Completed | 83 | 83
Not Completed | 16 | 15
Period: Follow-up >1 to <2 Years
Arm/Group | Soy Isoflavones | Placebo
Started | 83 | 83
Completed | 68 | 67
Not Completed | 15 | 16
Period: Follow-up 2 Years
Arm/Group | Soy Isoflavones | Placebo
Started | 68 | 67
Completed | 50 | 47
Not Completed | 18 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Soy Isoflavones | Placebo | Total
Number analyzed (Participants) | 99 | 98 | 197
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 99 | 98 | 197
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 98 | 197
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 51 | 39 | 90
  Not Hispanic or Latino | 48 | 59 | 107
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 99 | 98 | 197
FGBT% [Mean (Standard Deviation); unit: percentage of total breast] — Population: One placebo and 4 isoflavone participants had missing or unsatisfactory baseline images.
  percentage of total breast
    number analyzed (Participants) | 95 | 97 | 192
    (all) | 24.76 (14.54) | 23.86 (13.99) | 24.3 (14.23)

OUTCOME MEASURES:

1. Primary Outcome: Fibroglandular Tissue in Total Breast (FGBT%)
Description: Effects of 1 and 2 years of treatment with isoflavones on percent of changes in FGBT%.
Time Frame: baseline, and after year 1 and 2 of supplementation
Population: Subjects with at least 1 treatment image.
Measure: Mean (Standard Deviation); unit: percentage of total breast tissue
Arm/Group | Soy Isoflavones | Placebo
Number analyzed (Participants) | 68 | 67
percentage of total breast tissue
  Baseline | 24.94 (14.11) | 25.34 (14.93)
  Year 1: number analyzed (Participants) | 65 | 63
  Year 1 | 24.03 (15.34) | 25.82 (14.72)
  Year 2: number analyzed (Participants) | 50 | 49
  Year 2 | 23.14 (14.58) | 25.36 (13.38)
Statistical Analysis 1: Comparison: Soy Isoflavones vs Placebo; (FGBT% at 1 year of treatment minus FGBT% at baseline) divided by FGBT% at baseline; Test type: Other; p = 0.071, t-test, 2 sided
Statistical Analysis 2: Comparison: Soy Isoflavones vs Placebo; (FGBT% at 2 year of treatment minus FGBT% at baseline) divided by FGBT% at baseline; Test type: Other; p = 0.080, t-test, 2 sided
Statistical Analysis 3: Comparison: Soy Isoflavones vs Placebo; Intention to treat; Test type: Other; p = 0.019, Regression, Linear; Mixed model; Slope = -0.107, Standard Error of Mean 0.045 — slope for interaction of treatment and time, placebo was the reference group; square root transformed outcome

2. Primary Outcome: Breast Density by Mammography
Description: Area of FGBT in mammogram. The timepoints were combined and summed.
Time Frame: baseline, and after year 1 and 2 of supplementation
Population: Three Soy Isoflavones participants had missing mammograms.
Measure: Mean (Standard Deviation); unit: percentage of total breast
Arm/Group | Soy Isoflavones | Placebo
Number analyzed (Participants) | 96 | 98
percentage of total breast | 27.7 (11.62) | 26.73 (10.83)

3. Secondary Outcome: Bone Mineral Density
Description: Bone mineral density of hip, spine and whole body bone mineral density as measured by dual x-ray absorptiometry. The timepoints were combined and summed.
Time Frame: one and two years after dietary supplement
Population: Intention to treat participants. Two placebo and one isoflavone subjects had breast images but no DXA tests.
Measure: Mean (Standard Deviation); unit: g/cm^2
Arm/Group | Soy Isoflavones | Placebo
Number analyzed (Participants) | 98 | 96
g/cm^2
  Hip bone mineral density | 1.01 (0.12) | 1.00 (0.13)
  Spine bone mineral density | 1.06 (0.11) | 1.06 (0.11)
  Whole body bone mineral density | 1.08 (0.09) | 1.07 (0.09)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Soy Isoflavones | Placebo
All-Cause Mortality (participants affected / at risk) | 0/99 | 0/98
Serious Adverse Events (participants affected / at risk) | 0/99 | 0/98
Other Adverse Events (participants affected / at risk) | 1/99 | 6/98
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Soy Isoflavones (N=99) | Placebo (N=98)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 6
Presynocopy (Nervous system disorders) | 0 | 1
Hives (Skin and subcutaneous tissue disorders) | 0 | 1
Ear Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Lower Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 1
uterus, cervix, cyst and polyp in cervix (Reproductive system and breast disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-07-07): https://cdn.clinicaltrials.gov/large-docs/90/NCT00204490/Prot_SAP_000.pdf